CLINICAL TRIAL: NCT04134884
Title: A Phase I Study of ASTX727 Plus Talazoparib in Patients With Triple Negative or Hormone Resistant/ Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Metastatic Breast Cancer
Brief Title: Study of ASTX727 Plus Talazoparib in Patients With Triple Negative or Hormone Resistant/HER2-negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kathy Miller (Other)
Collaborators: Pfizer (Industry); Astex Pharmaceuticals, Inc. (Industry); Van Andel Institute Stand Up to Cancer Team (Unknown)
Responsible Party: Sponsor-Investigator, Kathy Miller, Ballvé-Lantero Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCC-0684
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer; Triple Negative Breast Cancer; Hormone Receptor Positive Tumor
Keywords: Breast Cancer; Phase 1
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — talazoparib; decitabine and cedazuridine drug combination

STUDY DESIGN:
Intervention Model Description: The dose escalation phase will begin by enrolling 3 patients to the cohort 1 dose level. Patients will be observed for 28 days or one cycle of therapy for dose limiting toxicity (DLT).
  If 0 of 3 patients experience a DLT, the study will proceed to cohort 2. If 1 patient experiences a DLT, 3 additional patients will be enrolled into cohort 1. If 1 of 6 patients experience a DLT, the study will proceed to the cohort 2 dose level. If > 2/3 or 2/6 patients in cohort 1 experience DLT, we will de-escalate to cohort -1. Identical DLT evaluation and dose escalation/de-escalation decision rules will be used in subsequent cohorts. A total of 6 patients will be treated at the highest dose level achieved to ensure that 6 patients have been treated at the proposed maximum tolerated dose before proceeding to the expansion cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASTX727 + Talazoparib (Experimental)
  Interventions: Drug: Talazoparib; Drug: ASTX727

INTERVENTIONS:
Drug: Talazoparib — Talazoparib will be taken on days 4-21, 6-21 or 1-21 at a dose level of 0.25, 0.5, 0.75 or 1.0 mg depending on cohort assignment
Drug: ASTX727 — ASTX727 will be taken on days 1 and 3, days 1,3,5 or days 1 through 5 of the 28 day cycle at doses of 10 mg:100 mg or 15 mg:100 mg depending on cohort assignment

SUMMARY:
This is a Phase I study to test the safety of a combination of ASTX727 with talazoparib in patients with triple negative breast cancer or hormone resistant/HER2-negative metastatic breast cancer

DETAILED DESCRIPTION:
The phase I portion will use a traditional 3 + 3 design and standard definitions of DLT based on toxicity experienced during the first cycle of therapy. Patients with triple negative breast cancer (TNBC) and hormone resistant/HER2 negative (HRBC) metastatic disease will be enrolled and analyzed together during the dose escalation cohorts. Once the maximum tolerated dose is determined, we will enroll a small expansion cohort to further characterize safety and provide preliminary efficacy estimates.The expansion cohort will be limited to 14 patients; 7 with TNBC and 7 with HRBC. The dose level selected for expansion will be based on the totality of the data available including toxicity during the DLT evaluation period, toxicity during subsequent cycles, and correlative results.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Locally recurrent (not amenable to local therapy with curative intent) or metastatic breast cancer

   1. Patients with triple negative breast cancer must have received at least one prior chemotherapy regimen for metastatic disease.
   2. Patients with hormone-positive, HER2-negative disease must have received treatment with and progressed on at least one prior endocrine therapy including a CDK4/6 inhibitor in the metastatic setting.
4. Measurable or evaluable disease based on RECIST 1.1 criteria.
5. Only subjects who have disease amenable to biopsy will be asked to consent to serial tumor biopsies. Consent for biopsy is not required for participation.

   a. NOTE: If no amendable disease is present at the time of biopsy, subjects may continue participation in the study and further study specific biopsies will not be required.
6. Eastern Cooperative Oncology Group Performance Status 0 or 1
7. Patients with treated, asymptomatic central nervous system (CNS) disease may participate if the patient is > 4 weeks from completion of CNS therapy (radiation and/or surgery), is clinically stable at the time of study entry, and is receiving a stable or decreasing dose of corticosteroid therapy. Brain MRI or head CT is required at screening for patients with known brain metastases.
8. Adequate organ function as indicated by:

   1. Total bilirubin </= ULN (upper limit of normal) (except in patients with documented Gilbert's disease, who must have a total bilirubin </= 3.0 mg/dL)
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 3.0 x ULN (</= 1.5-3.0 x baseline if baseline is abnormal)
   3. Calculated creatinine clearance of >/= 60 mL/min using the Cockcroft-Gault formula
   4. Absolute neutrophil count (ANC) >/= 1.5 K/mm3
   5. Platelets >/= 100 K/mm3
   6. Hemoglobin (Hgb) >/= 9.0 g/dL
9. Women of childbearing potential must have a negative pregnancy test within 14 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

   1. Has undergone a hysterectomy or bilateral oophorectomy; or
   2. Has been naturally amenorrheic for at least 24 consecutive months.
10. Women of childbearing potential and men must agree to use effective contraception throughout the study and for 7 months after the last study treatment. Note: Acceptable methods of birth control include abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections).

Exclusion Criteria:

1. Prior treatment with decitabine, guadecitabine or other known DNA Methyltransferase inhibitors (DNMTis)
2. Prior treatment with talazoparib or other known PARPi (poly(ADP-ribose polymeras inhibitor)
3. Known deleterious breast cancer susceptibility gene (BRCA) mutation. Patients with BRCA variants of unknown significance (VUS) or who have not had germline genetic testing may participate.
4. Active or symptomatic CNS disease
5. Patients with HER2+ disease

   * HER2 will be considered positive if scored 3+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of > 2.0 or > 6 total HER2 gene copies per cell.
6. Patients with active malignancy other than breast cancer. Patients with prior malignancies without recurrence after standard treatment will not be excluded
7. Chemotherapy within 3 weeks of registration
8. Radiation therapy within 2 weeks of registration
9. Hormone therapy within 2 weeks of registration
10. Patients requiring ongoing therapy with strong P-gp inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Safety of ASTX727 plus talazoparib using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0 | through study completion i.e up to 1 year
Rate of dose limiting toxicity | 28 days
  rate of dose limiting toxicity will be assessed during cycle 1 (28 days) in patients enrolled during the dose escalation phase

SECONDARY OUTCOMES:
Overall response rate | through study completion (i.e. up to 1 year)
Clinical benefit response for triple negative disease subjects | 18 weeks
  clinical benefit response defined as complete response, partial response, or stable disease
Clinical benefit response for hormone receptor positive/ HER2 negative subjects | 24 weeks
  clinical benefit response defined as complete response, partial response, or stable disease
Progression free survival in all enrolled subjects | through study completion (i.e. up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina